CLINICAL TRIAL: NCT06989281
Title: Randomized Encouragement Trial to Evaluate the Implementation and Effectiveness of a Lifestyle Medicine Clinic in Primary Care
Brief Title: Evaluation of a Primary Care Based Lifestyle Medicine Clinic at UAB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Drew Sayer, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-300013918
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Quality Improvement Project; Implementation; Clinical Effectiveness; Encouragement Design
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This QI project uses a randomized encouragement trial design. All patients of the UAB Family and Community Medicine Clinic will have access to the FLOW lifestyle medicine clinic via program brochures placed in the clinic and/or direct referral from their healthcare providers. Some patients (i.e., Encouraged condition) will be randomly assigned to receive extra encouragement to consider enrolling in the FLOW lifestyle medicine clinic. Because all patients have access to the clinic, the intervention is minimal risk, and the findings are specific to the UAB Medicine Health System, this project is being conducted without obtaining patient consent (non-human subjects research).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encouraged to Enroll in FLOW (Experimental): Patients randomized to this condition receive extra encouragement to consider enrolling in the FLOW lifestyle medicine clinic. This encouragement includes the addition of 2 questions added to their patients' pre-visit intake process regarding their interest in making healthy lifestyle changes to improve their cardiometabolic health. If affirmative, the Certified Medical Assistant will provide the patient with a FLOW brochure and make a note for the provider to follow-up with the patient and consider referral to the FLOW clinic.
  Interventions: Behavioral: FLOW Lifestyle Medicine Clinic
- Not Encouraged to Enroll in FLOW (Active Comparator): Patients randomized to this condition do not receive extra encouragement to enroll in the FLOW lifestyle medicine clinic. They are still able to access to the FLOW clinic via brochures placed in the waiting area and exam rooms or direct referral by their healthcare provider (without having been "encouraged.")
  Interventions: Behavioral: FLOW Lifestyle Medicine Clinic

INTERVENTIONS:
Behavioral: FLOW Lifestyle Medicine Clinic — The FLOW Lifestyle Medicine Clinic is a 12-month multidisciplinary program for improving obesity and obesity-related chronic conditions. FLOW is an evidence-based program that aligns with USPSTF recommendations for intensive behavioral counseling for obesity and cardiovascular disease risk reduction. There are at least 12 clinician/patient encounters in the FLOW clinic over 12 months including 6 with a registered dietitian and 6 with a FLOW physician. Behavioral Health assessments and visits are also offered as part of FLOW but are optional.

SUMMARY:
This is a randomized quality improvement project (i.e., not a research study) that will test the implementation and effectiveness of a lifestyle medicine clinic at the University of Alabama at Birmingham.

DETAILED DESCRIPTION:
This is a randomized quality improvement project that has received a non-human subjects research determination from the IRB at the University of Alabama at Birmingham. This study will use a randomized encouragement trial design to test whether a lifestyle medicine clinic at UAB (FLOW: Fitness, Lifestyle, and Optimum Wellness) is implementable and effective for improving cardiometabolic health (e.g., body weight, body composition, blood pressure, blood glucose, and blood lipids). Only patients of the UAB Family and Community Clinic are included in this project (i.e., no outside recruitment/enrollment).

ELIGIBILITY:
Inclusion Criteria:

* Current patient of the UAB Family & Community Medicine Clinic
* BMI: greater than or equal to 25 kg/m2
* Previous diagnosis of at least one of the following conditions:
* prediabetes or type 2 diabetes
* prehypertension or hypertension
* dyslipidemia

Exclusion Criteria:

* Not a current patient of the UAB Family & Community Medicine Clinic

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Referral | Baseline
  Comparison of rates of referral to the FLOW clinic between the Encouraged and Not Encouraged conditions.
Rate of Enrollment | Baseline
  Comparison of rates of enrollment in the FLOW clinic between the Encouraged and Not Encouraged conditions.

SECONDARY OUTCOMES:
ITT Estimand, Change in Body Weight | Baseline and 12 months
  A comparison body weight changes occurring over 12 months between patients assigned to Encouraged vs. Not Encouraged.
ITT Estimand, Change in Composite Cardiometabolic Health | Baseline to Month 12
  A comparison of changes in cardiometabolic health occurring over 12 months between patients assigned to Encouraged vs. Not Encouraged. The composite score is derived from values for body weight, percentage body fat, blood pressure, clinical labs, fitness tests, and questionnaires.
Complier Average Causal Effect, Change in Body Weight | Baseline and 12 months
  A comparison body weight changes occurring over 12 months between patients who enrolled vs. did not enroll in FLOW regardless of whether they were assigned to Encouraged or Not Encouraged.
Complier Average Causal Effect, Change in Composite Cardiometabolic Health | Baseline to Month 12
  A comparison changes in cardiometabolic health occurring over 12 months between patients who enrolled vs. did not enroll in FLOW regardless of whether they were assigned to Encouraged or Not Encouraged. The composite score is derived from values for body weight, percentage body fat, blood pressure, clinical labs, fitness tests, and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Drew Sayer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This project is a quality improvement project intended for improving obesity and obesity related cardiometabolic health among UAB patients. Because this project is not "research" (i.e., contributing to generalizable knowledge), we do not believe it is appropriate to share IDP with outside investigators.